CLINICAL TRIAL: NCT01890408
Title: Continuous Preperitoneal Infusion of Ropivacaine After Open Liver Resection: Effect on Post-operative Recovery and Morbidity
Acronym: ROPIHEP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: promoter decision
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P111101
Record Dates: First submitted 2013-06-14; First posted 2013-07-01 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Laparotomy; Hepatic Resection
Keywords: Laparotomy; Hepatic resection; continuous wound catheter analgesia; morphine; post operative recovery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ropivacaine (Experimental): patients scheduled to undergo open liver resection Age > 18 years Free from pain in preoperative period
  Interventions: Drug: wound infusion ropivacaine
- placebo (Placebo Comparator): patients scheduled to undergo open liver resection Age > 18 years Free from pain in preoperative period

INTERVENTIONS:
Drug: wound infusion ropivacaine — Laparotomy Hepatic surgery :
  Bolu of 10 ml de ropivacaine 0,2% + infusion with elastomeric pump with ropivacaine 0,2% at a 10ml/h during 48 hours.
  Arms: ropivacaine

SUMMARY:
Intravenous morphine Patient-Controlled analgesia is gold standard on post - operative liver resection. But, opioids tend to be ineffective for pain that is associated with movement and have significant short-term side effects including nausea, vomiting, sedation, pruritus, constipation, urinary, retention, and respiratory depression, which are factors that often hinder a patient's recovery. Prospective randomized trials has found continuous wound catheter analgesia as an accepted alternative to IV morphine PCA.

The researchers will investigate whether ropivacaine, administered through a wound catheter placed by the surgeon, will reduce morbidity and provide a better recovery.

DETAILED DESCRIPTION:
This study is a prospective, double blind, randomized study. Subjects will be randomized using a computer-generated table of random numbers into 2 groups. The patients scheduled to undergo open liver resection will be randomly allocated to receive a continuous wound infusion of either 0.2% ropivacaine (ropivacaine group A) or 0.9% saline (control group B). The patients will be thereafter randomly assigned to receive through the catheter either 0.2% ropivacaine (study group) (10-ml bolus followed by an infusion of 10 ml/h during 48 h) or the same protocol with 0.9% NaCl (control group), thanks to a elastomeric pump (500ml), set to deliver a 10-ml/h connected with the catheter. In addition, all patients will receive patient-controlled intravenous morphine analgesia. The primary endpoint : the opioid-related symptom distress scale (SDS) will be performed at 48 hours after surgery. Secondary endpoints will be pain intensity on a visual analog scale at rest, and on coughing, morphine consumption, respiratory dysfunction, transit recovery and side effects at 48 hours, 5 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Scheduled for open hepatic resection
* Patients must be able to understand the IV morphine PCA
* Written informed consent
* Free from pain in preoperative period

Exclusion Criteria:

* Age < 18 years
* Severe hepatic
* Renal impairment
* Pregnancy or lactation
* Allergy to one of the specific drugs under study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
the opioid-related symptom distress scale (SDS) | 48 h postoperatively

SECONDARY OUTCOMES:
Diaphragmatic function | 48 h, 5 days postoperatively and discharge
  Sniff-test and Peak-flow
total morphine consumption | 48 h, 5 days postoperatively and discharge
Recovery after surgery | 48 h, 5 days postoperatively and discharge
  It is defined as the time to first flatus and recovery of bowel activity after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Thibault Camus, Dr, Principal Investigator — Assistance Publique
Locations (1):
- Département anesthésie-réanimation, Paris, France